CLINICAL TRIAL: NCT02383199
Title: Polypropylene Mesh in Prolapse Surgery; Long-term Outcome and Complications.
Brief Title: Polypropylene Mesh in Prolapse Surgery
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 134/2013
Record Dates: First submitted 2015-02-02; First posted 2015-03-09 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to report the long-term objective and subjective outcome after prolapse surgery with polypropylene mesh. The complications and the effect of the learning curve of the surgeons to the outcome is also reported.

ELIGIBILITY:
195 first patients with pelvic organ prolapse operated on using polypropylene mesh

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 195 first patients with pelvic organ prolapse operated on a in Turku University Hospital using polypropylene mesh
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Subjective outcome with validated questionnaires | 7 years
  Validated questionnaires

SECONDARY OUTCOMES:
Objective outcome: anatomic outcome with Pelvic Organ Prolapse Quantification (POP-Q) system | 7 years
Number of patients with adverse events and reoperations. | 7 years
  POP-Q

CONTACTS AND LOCATIONS:
Overall Officials: Pia Heinonen, MD, Principal Investigator — Turku university hospital, Department of gynecology and obsteterics, Turku, Finland':'